CLINICAL TRIAL: NCT03136991
Title: A Phase I, Randomized, Single-blind, Placebo-controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD4831 After Multiple Ascending Dose Administration to Healthy Male Subjects
Brief Title: A Phase I, Safety Tolerability and Pharmacokinetics of AZD4831 to Treat Cardiovascular Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D6580C00004
Record Dates: First submitted 2017-04-27; First posted 2017-05-02 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Cardiovascular Disease
Keywords: Oral myeloperoxidase inhibitor
MeSH Terms: conditions — Cardiovascular Diseases | interventions — AZD4831

STUDY DESIGN:
Intervention Model Description: This study will be a randomized, single-blind (site personnel to remain blinded until SRC meeting), placebo-controlled, MAD, sequential group design study in healthy male subjects, performed at a single study center. Up to 60 healthy male subjects aged 18 to 50 years (inclusive) are planned to be investigated in 4 cohorts, but up to 6 cohorts may be included if the SRC considers it necessary to repeat a dose level or if additional dose levels are required.
  Up to 10 subjects will participate in each cohort. Within each cohort 8 subjects will be randomly assigned to receive AZD4831 and 2 subjects to receive placebo. AZD4831 or placebo will be administered once daily for a period of 10 days. It is anticipated this will be sufficient to achieve and maintain steady state PK profiles for several days, permitting evaluation of the safety and tolerability of multiple dose administrations at steady state. The subjects will stay at the study center during the whole dosing period and until 48h
Who Masked: Participant
Masking Description: This study will be a randomized, single-blind (site personnel to remain blinded until SRC meeting), placebo-controlled, MAD, sequential group design study in healthy male subjects, performed at a single study center.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Active Comparator): Participants will receive AZD4831 5 mg/placebo oral suspension.
  Interventions: Drug: AZD4831; Drug: Placebo
- Cohort 2 (Active Comparator): Participants will receive AZD4831 (Additional dose 1)/placebo oral suspension.
  Interventions: Drug: AZD4831; Drug: Placebo
- Cohort 3 (Active Comparator): Participants will receive AZD4831 (Additional dose 2)/placebo oral suspension.
  Interventions: Drug: AZD4831; Drug: Placebo
- Cohort 4 (Active Comparator): Participants will receive AZD4831 (Additional dose 3)/placebo oral suspension.
  Interventions: Drug: AZD4831; Drug: Placebo

INTERVENTIONS:
Drug: AZD4831 — Participants will receive AZD4831 once daily, orally, for a period of 10 days. Note: Additional doses (for cohorts 2,3&4) are provisional and could be adjusted based on the emerging data after the review of all available safety or other pertinent data from the previous dose by the Safety Review Committee (SRC).
Drug: Placebo — Participants will receive placebo matching the AZD4831 dose, once daily, orally, for a period of 10 days.

SUMMARY:
This is a Phase I study to investigate the safety and tolerability of AZD4831 in healthy male participants, conducted at a single center. The results from this study will form the basis for decisions on future studies. Another purpose of this dose escalation study is to find out the right dose of the experimental drug to be given to study participants in future studies. Even though there were no harmful effects seen in the animals tested, investigator does not know what side effects the experimental drug might cause in humans. However, site personnel managing the study participants will be blinded to the extent possible and as long as possible to minimize any impact on data collection. Study participants will be blinded to treatment allocation.

The study will be conducted in healthy participants to avoid interference from disease processes or other drugs.

The participants will stay at the study center during the whole dosing period and until 48 hours post final dose.

DETAILED DESCRIPTION:
This is a Phase I study to investigate the safety and tolerability of AZD4831 in healthy male participants, conducted at a single center.The results from this study will form the basis for decisions on future studies. Another purpose of this dose escalation study is to find out the right dose of the experimental drug to be given to study participants in future studies. The study will be conducted in healthy participants to avoid interference from disease processes or other drugs. The participants will stay at the study center during the whole dosing period and until 48 hours post final dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male participants aged 18 to 50 years (inclusive at Screening) with suitable veins for cannulation or repeated venipuncture.
* Have a BMI between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
* History or presence of gastrointestinal (GI), hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Presence of infection(s) (particularly fungal infection), as judged by the Investigator.
* History or current thyroid disease.
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP.
* Any clinically significant abnormalities in biochemistry, hematology, or urinalysis results, as judged by the Investigator at Screening and/or Day 1, including

  1. Alanine aminotransferase (ALT) not within normal range;
  2. Aspartate aminotransferase (AST) not within normal range;
  3. Creatinine not within normal range;
  4. White blood cell (WBC) not within normal range;
  5. Hemoglobin not within normal range; and
  6. Estimated Glomerular Filtration Rate (eGFR) not within normal range.
* Any positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody and human immunodeficiency virus (HIV) type 1 and 2.
* Abnormal vital signs, after 10 minutes supine rest, at Screening and/or Day 1, defined as any of the following:

  1. Systolic BP (SBP) < 90 mmHg or ≥ 140 mmHg
  2. Diastolic BP (DBP) < 50 mmHg or ≥ 90 mmHg
  3. Pulse < 45 or > 85 beats per minute (bpm)
* Persistent or intermittent complete bundle branch block, incomplete bundle branch block, or interventricular conduction delay with QRS > 110 ms. Participants with QRS > 110 ms but < 115 ms are acceptable if there is no evidence of, for example, ventricular hypertrophy or pre-excitation at Screening and/or Day 1.
* Electrocardiogram findings suggesting a metabolic or other non-cardiac condition that may confound interpretation of serial changes (such as hypokalemia) at Screening and/or Day 1.
* Use of any prescribed or non-prescribed medication (other than paracetamol/acetaminophen), including antacids, analgesics, herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks before the first administration of IMP or longer if the medication has a long half-life.
* Plasma donation within 1 month of Screening or any blood donation/blood loss > 500 mL during the 3 months before Screening.
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of IMP in this study. The period of exclusion begins 3 months after the final dose or 1 month after the last visit whichever is the longest.
* Vulnerable participants, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy male participants aged 18 to 50 years (inclusive at Screening) with suitable veins for cannulation or repeated venipuncture.
  Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive
Enrollment: 38 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-11-22 (Actual); Study Completion 2017-11-22 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | From screening (Day -28 to Day -2) until final follow-up (Day 24)
  An AE is the development of an undesirable medical condition or the deterioration of a preexisting medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. An undesirable medical condition can be symptoms (e.g., nausea, chest pain), signs (e.g., tachycardia, enlarged liver) or the abnormal results of an investigation (e.g., laboratory findings, ECG).
Systolic Blood pressure | At screening (Day-28 to Day-2), Day -1, treatment period (Day 1, Day 10 and Day 12) and final follow-up (Day 24)
  Base line Systolic blood pressure (in mmHg) will be measured at the pre-dose assessment on Day 1. Assessment in treatment period on Day 1 at 0.5, 1, 2, 3, 4, 6, 8 and 12 hours post-dose. On Day 10 at Pre-dose and 12 hours post-dose. On Day 12 at 48 hours post last dose. Measurements will be collected after the subject had rested in the supine position for at least 10 minutes.
Twelve lead safety electrocardiography (ECG) | At screening (Day-28 to Day-2), treatment period (Day 1 to Day 12), and final follow-up period (Day 24)
  A 12-lead ECG will be performed on Days 1, 2, 3, 6, 10 and 11: (collected at end of dECG recording) and any additional required by PI on Days 4, 5, 7 to 9 at Pre dose and at discharge on Day 12, plus any additional required by PI. A 12-lead ECG will be obtained after the subject rested in the supine position for at least 10 minutes (For time-points coinciding with dECG measurements, a paper printout of the Schiller Cardiovit CS-200 recorder[ at the end of the 5- or 10-minute dECG recording], will be used and the result recorded. For time-points not coinciding with dECG measurements, the ECG recording will be directly recorded in ClinBase™ using ClinBase™ Cardiosoft™).
Twelve lead digital electrocardiography (dECG) | Treatment Period (Day 1 to Day 12)
  12-lead continuous dECGs will be recorded over at least 5 minutes on Day 1, 2, 3, 6, 10, 11 & 12. The AstraZeneca (AZ) ECG Centre will perform the digital ECG (dECG) analysis in this study, using the EClysis© system, version 3.4, or higher. At protocol-indicated time points, 12-lead continuous dECG will be recorded over at least 5 minutes with the Schiller Cardiovit CS-200 recorder (Schiller AG, Baar, Switzerland) and transmitted to the AZ central dECG repository, according to AZ ECG Centre´s standard procedures for settings, recording and transmission of dECGs. Time-points for dECG may be adjusted according to emerging PK data. All ECG recordings will be preceded by a 10-minute controlled rest period.
Telemetry | At Day -1 and treatment period (Day 1 and Day 10)
  A 2-lead real-time telemetry ECG will be performed for at least 4 hours on Day -1 and from 30 minutes pre-dose until 24 hours post dose. The telemetry monitoring system will be reviewed by the Investigator or research nurse and paper printouts of any clinically important events will be stored as source data.
Hematology | At screening (Day -28 to Day -2), Day -1, treatment period (Day 1, Day 10 and Day 12), final follow-up (Day 24)
  Number of clinically relevant new findings or worsening of a pre-existing findings as assessed by Haematology: Hematocrit (HCT), hemoglobin (Hb), red blood cell count (RBC), mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), white blood cell count (WBC), differential blood count (neutrophils, lymphocytes, monocytes, eosinophils and basophils), reticulocytes absolute count, and platelets. Assessments will be performed during treatment period on Day 1 at pre-dose, Day 10 at pre-dose and on Day 12 at 48 hour post final dose before check-out.
Physical examination | At screening (Day-28 to Day-2), Day -1, treatment period (Day 2 and Day 12), and final follow-up period (Day 24)
  A full physical examination will include the assessment of the following: general appearance, skin, cardiovascular, respiratory, abdomen, head, and neck (including ears, eyes, nose, and throat), lymph nodes, thyroid, musculoskeletal and neurological systems. A full physical examination will be performed at screening visit and at final follow-up visit (Day 24).
  A brief physical examination will include assessment of the following: general appearance, skin, cardiovascular system, respiratory and abdomen. A brief physical examination will performed at Day-1, treatment period (Day 1 to Day12) on Day 2: 24 h post first dose, and on Day 12: 48 h post final dose before check-out.
Diastolic blood pressure | At screening (Day-28 to Day-2), Day -1, treatment period (Day 1, Day 10 and Day 12) and final follow-up (Day 24)
  Base line diastolic blood pressure (in mmHg) will be measured at the pre-dose assessment on Day 1. Assessment in treatment period on Day 1 at 0.5, 1, 2, 3, 4, 6, 8 and 12 hours post-dose. On Day 10 at Pre-dose and 12 hours post-dose. On Day 12 at 48 hours post last dose. Measurements will be collected after the subject had rested in the supine position for at least 10 minutes.
Pulse rate | At screening (Day-28 to Day-2), Day -1, treatment period (Day 1, Day 10 and Day 12) and final follow-up (Day 24)
  Base line pulse rate (in beats per minute (bpm)) will be measured at the pre-dose assessment on Day 1. Assessment in treatment period on Day 1 at 0.5, 1, 2, 3, 4, 6, 8 and 12 hours post-dose. On Day 10 at Pre-dose and 12 hours post-dose. On Day 12 at 48 hours post last dose. Measurements will be collected after the subject had rested in the supine position for at least 10 minutes.
Oral body temperature | At screening (Day-28 to Day-2), Day-1, treatment period (Day 1 and Day 10 pre-dose)
  Oral temperature will be collected after the subject has rested in the supine position for at least 10 minutes.
Biochemistry | At screening (Day -28 to Day -2), Day -1, treatment period (Day 1 pre-dose, Day 10 pre-dose and Day 12 - 48 hours post final dose before check-out) and final follow-up (Day 24)
  Number of clinically relevant new findings or worsening of a pre-existing findings as assessed by serum biochemistry. Electrolytes: Sodium, potassium, calcium, and phosphate. Enzymes: Aspartate aminotransferase (AST), alanine aminotransferase (ALT), Alkaline phosphatase (ALP), gamma glutamyl transpeptidase (GGT), high-sensitivity C-reactive protein (hs-CRP). Substrates: Glucose (fasting), creatinine, total bilirubin, unconjugated bilirubin, conjugated bilirubin, albumin, and urea.
  For serum creatinine testing, blood samples will be collected on Day -1, pre-dose on Day 1, Day 5 and Day 10, follow-up (Day 14, Day 16 and Day 20) and final follow-up (Day 24)
Urinalysis | At Day -1, treatment period (pre-dose - Day 1, day 5 and Day 10), follow-up (Day 14, day 16 and Day 20) and final follow-up (Day 24)
  Dipstick analysis will be performed at the centre and includes: glucose, creatinine, protein, and blood.
Microscopy | At Day -1, treatment period (pre-dose - Day 1, day 5 and Day 10), follow-up (Day 14, day 16 and Day 20) and final follow-up (Day 24)
  Microscopy (RBC, WBC and casts [Hyaline, Granular and Cellular]) by thermodilatometry (TDL) may be performed at additional urinalysis time points if clinically relevant abnormalities are detected (positive result for protein or blood in dipstick).
Immunology | At Day -1, treatment period (Day 1 to Day 12), follow-up visits
  Number of clinically relevant new findings or worsening of a pre-existing findings as assessed by Immunology: Anti-neutrophil cytoplasmic antibodies (ANCA - a & p) testing and complements (C3a, C5a & Bb). ANCA serum testing will be performed on samples collected on Day -1, pre-dose on Day 1 and on Day 10 and at the final Follow-up Visit (Day 24). Complement testing will be performed on samples collected on Day -1, pre-dose on Day 1, Day 5 and Day 10, follow-up (Day 14, Day 16 and Day 20) and final follow-up (Day 24)

SECONDARY OUTCOMES:
Observed maximum concentration, taken directly from the individual concentration-time curve(Cmax) of AZD4831 and its metabolites | Day 1 and Day 10
  Observed maximum concentration.
Time to reach maximum concentration, taken directly from the individual concentration-time curve (tmax) of AZD4831 | Day 1 to Day 10
  Time to reach maximum concentration.
Observed trough plasma concentration [measured concentration at the end of the dosing interval taken just prior to the next administration] (Ctrough) of AZD4831 | Day 2 to Day 10
  Observed trough plasma concentration.
Terminal half-life (t1/2λz), estimated as (ln2)/λz) of AZD4831 | Day 10
  Terminal elimination half-life.
Area under the plasma concentration-curve over 24 hours (AUCτ) of AZD4831 | Day 1 and Day 10
  Area under the plasma concentration over 24 hours.
Area under the plasma concentration-time curve over the dosing interval divided by the dose administered (AUCτ/D) of AZD4831 | Day 1 and Day 10
  Area under the plasma concentration-time curve over the dosing interval divided by the dose administered.
Observed maximum plasma concentration divided by the dose administered (Cmax/D) of AZD4831. | Day 1 and Day 10
  Observed maximum plasma concentration divided by the dose administered.
Apparent clearance for parent drug (CL/F) estimated as dose divided by AUCτ of AZD4831. | Day 10
  Apparent clearance for parent drug.
Mean Residence Time (MRT) | Day 10
  Mean Residence Time.
Apparent volume of distribution for parent drug at terminal phase(Vz/F)(extravascular administration), estimated by dividing the apparent clearance (CL/F) by λz of AZD4831. | Day 10
  Apparent volume of distribution for parent drug at terminal phase.
Accumulation ratio calculated as AUCτ Day 10/ AUCτ Day 1 (RacAUC) of AZD4831. | Day 10
  Accumulation ratio calculated as AUCτ Day 10/ AUCτ Day 1.
Accumulation ratio calculated as Cmax Day 10/ Cmax Day 1 (Rac Cmax) of AZD4831. | Day 10
  Accumulation ratio calculated as Cmax Day 10/ Cmax Day 1.
Amount of analyte excreted into the urine from time t1 to t2 (Ae(t1-t2)) of AZD4831. | Day 1 and Day 10
  Amount of analyte excreted into the urine.
Cumulative amount of analyte excreted at time t (Ae(0-t)) of AZD4831. | Day 1 and Day 10
  Cumulative amount of analyte excreted at time t.
Fraction of dose excreted unchanged into the urine from time t1 to t2, estimated by dividing Ae(t1-t2) by dose (fe(t1-t2)) of AZD4831. | Day 1 and Day 10
  Fraction of dose excreted unchanged into the urine.
Fraction of dose excreted unchanged into the urine from time zero to time t, estimated by dividing Ae(0-t) by dose (fe(0-t)) of AZD4831 | Day 1 and Day 10
  Fraction of dose excreted unchanged into the urine.
Renal clearance, estimated by dividing Ae(0-t) by AUC(0-t), using appropriate matching time t (CLR) of AZD4831. | Day 1 and Day 10
  Renal clearance.
Terminal rate constant, estimated by log-linear least-squares regression rate constant, estiamteed by log-linear least-squares (λz) | Day 10
  Terminal rate constant

CONTACTS AND LOCATIONS:
Overall Officials: David Han, MD, Principal Investigator — California Clinical Trials Medical Group 1560 East Chevy Chase Dr., Suite 140 Glendale, CA 91206
Locations (1):
- Research Site, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Undecided